CLINICAL TRIAL: NCT04010500
Title: Speech Performance of Rugby Players When Using Different Types of Mouthguard
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amy Liew (Other)
Responsible Party: Sponsor-Investigator, Amy Liew, Lecturer, Universiti Kebangsaan Malaysia Medical Centre
Organization: Universiti Kebangsaan Malaysia Medical Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UKMPPI/111/8/JEP-2018-278
Record Dates: First submitted 2019-06-28; First posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Speech
Keywords: dental trauma; rugby; mouthguard; speech; contact sports
MeSH Terms: conditions — Speech

STUDY DESIGN:
Intervention Model Description: The participants will articulate phonemes with plosive sounds (/p/, /b/, /d/ and /t/) for the following conditions in a pre-determined sequence: (i) not using mouthguard; (ii) using a 'boil and bite' mouthguard; and (iii) using a custom-fitted mouthguard. A washout interval of one hour will be implemented between conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rugby Players (Experimental)
  Interventions: Device: no mouthguard; Device: 'boil and bite' mouthguard; Device: custom-fitted mouthguard

INTERVENTIONS:
Device: no mouthguard — Control (not using mouthguard)
Device: 'boil and bite' mouthguard — KHZ058 Bicolor Mouth Guard (Shenzhen Kanghao Industrial Co. Ltd, China) will be immersed in a bowl of hot water (about 80 °C). After 50 seconds, the softened sheet will be fitted on the maxillary arch of the participant. The participant will then bite down to ensure the mouthguard stay firmly on the maxilla. After that, the mouthguard will be removed and immersed in cold water to retain its shape.
Device: custom-fitted mouthguard — The custom-fitted mouthguards will be constructed using the dual laminated technique with two layers of ethylene vinyl acetate (EVA) thermoplastic sheets (Dentsply International Raintree Essix, Court East Sarasota, USA).

SUMMARY:
Participation in contact sports is linked to an increased risk of dental injuries. To reduce the risk and severity of sports-related dental injuries, mouthguards are often recommended to be worn during training and competition. However, athletes often complain that they cannot talk properly when using mouthguards. It is hypothesized that speech performance differs when using different types of mouthguards. A group of female national rugby players will be asked to pronounce four Malay words with plosive sounds (/p/, /b/, /d/ and /t/) repeatedly in three conditions: (i) when not using any mouthguard, (ii) when using 'boil and bite' mouthguard, and (iii) when using custom-fitted mouthguard. The sounds will be recorded for spectrographic analysis. The difference in mean voice onset time between conditions will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* adult female aged 18 years old and older
* currently representing the nation and participating actively in rugby
* native speakers of Malay (national language)

Exclusion Criteria:

* did not play rugby within the last six months
* edentulism
* used a mouthguard, orthodontic appliance or removable prosthodontics appliance within the last six months
* known history of allergy to polymers
* medical problems (ASA classification 3 and above)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Mean voice onset time | Immediate
  The delay between the start of the speech sound and the beginning of vocal cord vibration (in millisecond)

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Kebangsaan Malaysia, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT04010500/Prot_SAP_000.pdf